CLINICAL TRIAL: NCT01613898
Title: Evaluation of Carotid IMT and Atherogenic Risk Factors in Patients With Cerebrotendinous Xanthomatosis
Acronym: CTX
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: SHEBA-09-7393-HC-CTIL
Record Dates: First submitted 2012-05-22; First posted 2012-06-07 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Cerebrotendinous Xanthomatosis (CTX)
Keywords: Cerebrotendinous xanthomatosis (CTX),; lipoprotein,atherosclerosis,; carotid artery intima-media thickness (cIMT).
MeSH Terms: conditions — Xanthomatosis, Cerebrotendinous; Atherosclerosis | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Lipid and lipoprotein profiles
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CTX Group
  Interventions: Biological: Blood tests

INTERVENTIONS:
Biological: Blood tests — Blood tests
  Other Names: CTX Group

SUMMARY:
The aim of the proposed study is to evaluate the risk for cardiovascular disease and 'atherogenic' features of the serum in CTX and to determine preclinical atherosclerosis. The study will include an extensive assessment of lipoprotein profile and carotid artery intima-media thickness (cIMT) measurement.

Lipid and lipoprotein profiles will include novel tests such as direct measurements of apolipoprotein A1,B,C2,C3 plasma levels, lipoprotein (a) levels, highly sensitive C-reactive protein levels and PLAC test that measures the levels of lipoprotein-associated phospholipase A2-a vascular-specific inflammatory enzyme implicated in the formation of atherosclerosis

DETAILED DESCRIPTION:
Protocol 09-2009 EVALUATION OF CAROTID IMT AND ATHEROGENIC RISK FACTORS IN PATIENTS WITH CEREBROTENDINOUS XANTHOMATOSIS

ABSTRACT Cerebrotendinous xanthomatosis (CTX) is a rare disease characterized by xanthomatous lesions in many tissues, mainly in the brain. Mutation in the gene of sterol 27-hydroxylase-an enzyme in bile acid synthesis causes CTX. The impaired synthesis of chenodeoxycholic acid from cholesterol results in elevated plasma and bile cholestanol.

The natural course of CTX is progressive neurologic deterioration from childhood through adulthood leading to diffuse damage of the central and peripheral nervous systems and eventually to death.

Cardiovascular involvement in CTX is probably high: different clinical manifestations of cardiovascular disease (CVD) were reported in 10.4% of patients with CTX. The precise mechanism of the atherosclerosis in CTX is unknown and may be related to cholestanol accumulation in the vascular subendothelial space.

Abnormalities in the lipoprotein profile were not described in the literature, and cholesterol levels are within normal limits in CTX. Extensive evaluation for CVD risk factors in the CTX patient group have not been conducted apart from a small number of publications.

The aim of the proposed study is to evaluate the risk for cardiovascular disease and 'atherogenic' features of the serum in CTX and to determine preclinical atherosclerosis. The study will include an extensive assessment of lipoprotein profile and carotid artery intima-media thickness (cIMT) measurement.

Lipid and lipoprotein profiles will include novel tests such as direct measurements of apolipoprotein A1,B,C2,C3 plasma levels, lipoprotein (a) levels, highly sensitive C-reactive protein levels and PLAC test that measures the levels of lipoprotein-associated phospholipase A2-a vascular-specific inflammatory enzyme implicated in the formation of atherosclerosis.

This would be the first attempt to conduct such an extensive evaluation in the CTX patients group.

Research Plan:

Study Design and Methods

Subjects The study population will constitute of all 17 CTX diagnosed patients that will be recruited from the CTX outpatient clinic at the Parkinson's disease and movement disorders Clinic in the Sagol Neuroscience Center, at the Chaim Sheba Medical Center. Patients will be contacted by phone and by mail and be invited to participate.

Control group will consist of age and gender matched healthy individuals. All patients or their legal guardians will sign an informed consent.

Detailed Plan of the Study

All study participants will undergo an evaluation that will include one clinic visit :

Visit 1

* A detailed medical history, including demographic data, past medical history, smoking history, use of medications, and family history of dyslipidemia and atherosclerotic cardiovascular disease.
* Physical examination including height and weight measurements, blood pressure, BMI, waist and hip circumference.
* Blood samples

  1. Fasting Lipid profile:

     Total cholesterol, HDL-cholesterol, direct LDL-cholesterol and Triglycerides (TG)
  2. Apolipoprotein profile:

  <!-- -->

  1. apolipoprotein A1
  2. apolipoprotein B
  3. apolipoprotein C2
  4. apolipoprotein C3

  c. lipoprotein (a) [Lp(a)] d. C-Reactive Protein -hsCRP e. Lipoprotein-associated Phospholipase A2 (Lp-PLA2) f. Apo E genotyping g. Plasma cholestanol level h. Fasting plasma glucose and Insulin
* 12 lead electrocardiogram (ECG)
* cIMT assessment.

Methods:

* Laboratory studies
* Blood samples will be taken after an overnight fast
* Total cholesterol, HDL-cholesterol and TG in plasma will be determined by colorimetric enzymatic procedures (Olympus, Ireland).
* Apolipoprotein A1, B, C2, C3 and Lp(a) serum concentrations will be determined by the immuno-turbidimetric procedure . (Olympus, Ireland).
* Direct LDL- will be determined by enzymatic color test. (Olympus, Ireland).
* HsCRP- will be determined by turbidimetric immunoassay(Olympus, Ireland)
* Lp-PLA2 (PLAC® Test) - The PLAC Test measures Lp-PLA2 (lipoprotein-associated phospholipase A2), a vascular-specific inflammatory enzyme implicated in the formation of rupture-prone plaque. Turbidimetric Immunoassay for the Quantitative Determination of Lp-PLA2 in Human Plasma (diaDexus, Inc. CA .USA) The Olympus AU 400 autoanalyzer will be used for all the above-mentioned measurements.
* Apo E genotyping- Apo E genotypes of genomic DNA from blood will be determined by a single nucleotide primer extension Elisa assay. (Pronto Diagnostics, Tel Aviv, Israel )
* Plasma cholestanol level- will be measured by high-performance liquid chromatography with ultraviolet detection (Halperin et al , ref 10 )
* Glucose -will be measured by the glucose oxidase method (Olympus AU2700, Hamburg, Germany).
* Insulin- will be measured by a chemiluminiscent immunometric method (Immulite 2000, Diagnostic Products Corporation, Los Angeles, CA).
* ECG-12 lead electrocardiogram will be done. (Mac 1100,GE medical systems, Germany)

Carotid artery Intima-media thickness : Patients will undergo a color-coded duplex examination of neck vessels using a 10MHz linear array ultrasound (Hitachi medical corporation, Tokyo, Japan). IMT will be evaluated on the common carotid arteries (CCAs) over ≈1.5 cm proximal to the flow divider, according to standardized guidelines. In brief, IMT will be measured at the thickest plaque-free point on the near and far walls with a specially designed computer program. CCA wall thickness will be defined as the mean of the maximum wall thickness of the near and far walls bilaterally. Ultrasound images of the distal 1 cm of the far wall of each common carotid artery will be obtained and compared with values from a normative data set (age and sex matched). Mean CIMT values from the far walls of the right and left common carotid arteries will be reported

ELIGIBILITY:
Inclusion Criteria:

* The study population will constitute of all 17 CTX diagnosed patients

Exclusion Criteria:

* Non CTX patients

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: PATIENTS WITH CEREBROTENDINOUS XANTHOMATOSIS
Sampling Method: Probability Sample
Enrollment: 17 (Estimated)
Dates: Start 2010-08; Primary Completion 2013-05 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Predisposition of CTX patients for pro-atherogenic features as evaluated by lipid and lipoproteins plasma profiles, and blood chemical assessment. Preclinical atherosclerosis in CTX patients as determined by Carotid artery Intima-media thickness 1. | 3 years
  The predisposition of the serum of CTX patients to be pro-atherogenic will be evaluated by detailed lipid and lipoproteins plasma profiles, and blood chemical assessment of specific inflammatory pro-atherogenenic features.
  IMT Presence of preclinical atherosclerosis will be determined by Carotid artery Intima-media thickness as a marker of risk for cardiovascular disease.

CONTACTS AND LOCATIONS:
Overall Officials: Hofit Cohen, MD, Principal Investigator — The Bert W. Strassburger Lipid Center
Locations (1):
- The Bert W. Strassburger Lipid Center, Tel Litwinsky, Israel